CLINICAL TRIAL: NCT07138378
Title: An Open-label, Randomized, Four-treatment, Four-period, Four-sequence, Single Dose, Crossover Study to Evaluate the Dose Adjusted Relative Bioavailability of Nilotinib Following the Oral Administration of Tasigna 200 mg Capsules, Tasigna 400 mg, XS003 (Nilotinib) Capsules 96mg and 192mg in Healthy, Adult Subjects Under Fasted Conditions
Brief Title: A Bioavailability Study of Nilotinib in Healthy, Adult, Human Subjects Under Fasted Conditions.
Acronym: XS003-11
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xspray Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: XS003-11
Record Dates: First submitted 2025-07-29; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — nilotinib

STUDY DESIGN:
Intervention Model Description: An open label, single-center, balanced, randomized, four-treatment, four-sequence, four-period, single dose, crossover, dose proportional study in healthy, adult, human subjects under fasting conditions.
Masking Description: This is an open label study. The bioanalytical personnel will be blinded to the randomization schedule until bioanalysis completed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tasigna 200 mg (Active Comparator): A single oral dose of Treatment Tasigna 200 mg
  Interventions: Drug: XS003 (nilotinib); Drug: Tasigna (nilotinib)
- Tasigna 400 mg (Active Comparator): A single oral dose of Treatment Tasigna 400 mg
  Interventions: Drug: XS003 (nilotinib); Drug: Tasigna (nilotinib)
- XS003 (nilotinib) 96mg (Experimental): A single oral dose of Treatment XS003 Capsules 2x48mg (96mg)
  Interventions: Drug: XS003 (nilotinib); Drug: Tasigna (nilotinib)
- XS003 (nilotinib) 192mg (Experimental): A single oral dose of Treatment XS003 Capsules 4x48mg (192mg)
  Interventions: Drug: XS003 (nilotinib); Drug: Tasigna (nilotinib)

INTERVENTIONS:
Drug: XS003 (nilotinib) — To evaluate the PK dose proportionality of Tasigna 200 mg versus Tasigna 400 mg and XS003 capsules 2x48mg (96mg) versus XS003 capsules 4x48mg (192mg).
Drug: Tasigna (nilotinib) — To evaluate the PK dose proportionality of Tasigna 200 mg versus Tasigna 400 mg and XS003 capsules 2x48mg (96mg) versus XS003 capsules 4x48mg (192mg).

SUMMARY:
An open label, single-center, balanced, randomized, four-treatment, four-sequence, four-period, single dose, crossover, comparative bioavailability study in healthy, adult, human subjects under fasteding conditions

DETAILED DESCRIPTION:
To evaluate the relative bioavailability of XS003 capsules 2x48mg (96mg) versus Tasigna 200 mg, and XS003 capsules 4x48mg versus Tasigna 400 mg after a single dose under fasted conditions in healthy, adult, human subjects.

ELIGIBILITY:
Inclusion Criteria:

A willing study participant to become eligible for the study must fulfill all of the below inclusion criteria:

* Healthy, human beings 18 and 45 years of age (both inclusive).
* Subjects weighing at least 50 kg, having a body mass index between 18.5 Kg/m2 and 29.9 Kg/m2 (both inclusive).
* Subject must be able to provide written informed consent with a detailed description of nature of the drug.
* Acceptable medical history, physical examination, ECG, laboratory investigations within 21 days prior to enrollment and chest X-ray (Valid for 180 days).
* Female subjects must meet one of the following criteria:

  * Physiological postmenopausal status, defined as the following.
  * Absence of menses for at least one year prior to the first study drug administration (without an alternative medical condition); and
  * FSH levels ≥40 mlU/mL at screening or
  * Surgical postmenopausal status, defined as the following.
  * Bilateral Oophorectomy and
  * Absence of menses for at least 90 days prior to the screening or
  * Post hysterectomy status
  * If postmenopausal and has an FSH of < 40 mlU/mL, but meets all other criteria in (i), (ii) or (iii) above as well as all the other inclusion criteria, screening estradiol serum level must be ≤ 150 pmol/L.

or

* iv.Surgically rendered non-childbearing potential by bilateral tubal ligation
* Must agree to use an adequate method of contraception. Subjects who are sexually active must use, with their partner, a condom AND one of the following methods of highly effective contraception from the time of IMP administration until 90 days after the last dose of IMP
* oral (except low-doselow dose gestagen (lynestrenol and norestisteron)), injectable or implanted hormonal contraceptives
* intrauterine device or system (e.g., progestin-releasing coil)
* vasectomized male (with appropriate post vasectomy documentation of the absence of sperm in the ejaculate)
* bilateral tubal occlusion or hysterectomy

  * Clinical laboratory values should be within the laboratory's stated normal range. If not within this range, they must be without clinical significance, as determined by the Investigator.
  * The subject is able to communicate meaningfully with study personnel and is anticipated to be able to comply fully with study procedures and must be willing and able to communicate and participate in the whole study.
  * Male subjects should not donate sperm during the study and for 90 days after the last administration of IMP.
  * Non-smokers .

Exclusion Criteria:

A willing study participant will be excluded from the study, if any of the below criteria is met:

* Systolic blood pressure less than 100 mm of Hg or more than 140 mm of Hg.
* Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg.
* Note: If vital signs are out-of-range, the investigator may obtain one additional reading so that up to 2 consecutive assessments are made within 1.00 hour with the subject seated quietly during the 5 minutes preceding the assessment.
* Body temperature less than 95.0 °F (35.0 °C) or more than 98.6°F (37.0°C).
* Radial Pulse rate less than 60/min or more than 100/min.
* History of hypersensitivity or idiosyncratic reaction to investigational drug product or any other related drugs.
* History of malignancy, cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, or psychiatric disease or disorder.
* Taken drugs that are substrates or inhibitors of P-glycoproteins in last 30 days prior to the check-in (see Appendix-5).
* History of hematological, malignant, and bleeding disorders.
* On anticoagulant therapy.
* History of hypokalemia, hypomagnesemia, or a history of cardiac disease.
* History of cholecystectomy or gall stones.
* History of any drug or alcohol abuse in the past 2 years.
* History of intake of strong CYP3A4 inhibitors (see Appendix-5) or inducers within
* 4 weeks prior to the check-in.
* History of intake of drugs known to prolong the QTc interval within 4 weeks prior to the check-in
* History of rare hereditary problems of galactose intolerance, severe lactase deficiency with a severe degree of intolerance to lactose-containing products, or of glucose-galactose malabsorption.
* A prolonged QTc interval (QTc greater than 450 msec demonstrated on ECG at Screening.
* Any clinically significant ECG abnormalities that, in the Investigator's opinion, would compromise the subject's safety.
* Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type).
* History or family history of long QT syndrome.
* Significant history or current evidence of risk factors for Torsade de Pointes (TdP).
* History of Gilbert syndrome.
* A history of difficulty with donating blood and having poor vein access.
* Male subjects with pregnant or lactating partners.
* Taking, or have taken, any prescribed or over-the-counter drug or herbal remedies, vitamins, or minerals and intake of any medication except caffeine, ranitidine, paracetamol, diclofenac sodium and ondansetron in the 30 days before check-in (other than up to 4 gr of paracetamol per day).
* Consumption of the xanthine containing food or beverages (like tea, coffee, chocolates, and flavored drinks) at least 48 hours before check-in of each period.
* Consumption of the grapefruit or grapefruit juice, pomegranate, or pomegranate juice, pomelo, starfruit, Seville oranges and St. John's Wort at least 14 days before check-in of each period.
* Consumption of tobacco containing products (including smoking cigarettes or chewing tobacco products), e-cigarettes and/or nicotine replacement products within 3 months prior to the check-in.
* Consumption of all kinds of alcoholic beverages from at least 48.00 hours prior to check-in.
* Difficulty in abstaining from all kinds of alcoholic beverages during entire study period.
* Difficulty in abstaining from the xanthine containing food or beverages (like tea, coffee, chocolates, and flavored drinks), grapefruit or grapefruit juice, pomelo, pomegranate, or pomegranate juice, pomelo, starfruit, Seville oranges and St. John's Wort during entire study period.
* Difficulty in abstaining from the smoking or chewing tobacco products during entire study period.
* Confirmed positive for drugs of abuse (benzodiazepines, tetrahydrocannabinol, amphetamine, cocaine, barbiturates, and morphine) on check-in of any period.
* Confirmed positive alcohol (breath) test on check-in of any period.
* Confirmed positive urine cotinine test on check-in of any period.
* Participated in any other clinical study or donated blood in last 90 days.
* Positive screens for serum hepatitis B surface antigen (HbsAg), hepatitis C antibody (HepC) or human immunodeficiency virus (HIV).
* Participated in contact sports or unaccustomed strenuous exercise in the 72 hours before check-in of any period.
* History of clinically significant allergy.
* History of allergy or sensitivity to nilotinib, or history of any food or drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
* Significant history or current evidence of chronic infectious disease, system disorders, organ dysfunction especially cardiovascular disorders (e.g., arterial vascular occlusive events), respiratory disorders, renal or hepatic disorders, diabetes, or obesity.
* Greater than the upper limit of normal values of Alkaline phosphatase (ALP), alanine transaminase (ALT), aspartate aminotransferase (AST) and total bilirubin.
* Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m2 at period-1
* check-in.
* Clinically significant hypokalemia, hypomagnesemia, or other electrolyte disorders.
* Clinically significant history or presence of gastrointestinal disease or history of malabsorption within the last year, as determined by the Investigator.
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* Confirmed positive pregnancy test (for females) on check-in of any period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Bioavailability (Peak Plasma Concentration (Cmax)) of XS003 versus Tasigna treatment | PK samples will be collected at pre-dose (0.00) and between 0.50 and 120.00 hours post dose
  To evaluate the relative bioavailability (Peak Plasma Concentration (Cmax)) of XS003 capsules 2x48mg (96mg) versus Tasigna 200 mg, and XS003 capsules 4x48mg versus Tasigna 400 mg after a single dose under fasted conditions in healthy, adult, human subjects.
Bioavailability (Area under the plasma concentration versus time curve (AUC)) of XS003 versus Tasigna treatment | PK samples will be collected at pre-dose (0.00) and between 0.50 and 120.00 hours post dose
  To evaluate the relative bioavailability (Area under the plasma concentration versus time curve (AUC)) of XS003 capsules 2x48mg (96mg) versus Tasigna 200 mg, and XS003 capsules 4x48mg versus Tasigna 400 mg after a single dose under fasted conditions in healthy, adult, human subjects.

SECONDARY OUTCOMES:
Safety (adverse events (AE)) of XS003 versus Tasigna treatment | From baseline up to 58 days
  To evaluate the safety and tolerability (adverse events (AE, i.e treatment and non-treatment related adverse events as assessed by CTCAE v4.0)) of Tasigna 200 mg, Tasigna 400 mg, XS003 Capsules 2x48mg (96mg) and 4x48mg (192mg) in healthy, adult, human subjects under fasted conditions.
Safety (electrokardiografi ECG)) of XS003 versus Tasigna treatment | From baseline up to 58 days
  To evaluate the safety and tolerability (electrokardiografi ECG QT Interval)) of Tasigna 200 mg, Tasigna 400 mg, XS003 Capsules 2x48mg (96mg) and 4x48mg (192mg) in healthy, adult, human subjects under fasted conditions

CONTACTS AND LOCATIONS:
Overall Officials: Maria Klockare, Study Director — Xspray Pharma
Locations (1):
- QPS Bioserve India Pvt Limited, Hyderabad, India

IPD SHARING:
Plan to Share IPD: No
N/A as this is a Bioavailibility study